CLINICAL TRIAL: NCT05304494
Title: Sentinel - Triaging Acute Breathlessness Using Multi-Modal Biomarkers
Status: Withdrawn | Type: Observational
Why Stopped: Limited resources
Sponsor: Sanome (Industry)
Responsible Party: Sponsor
Other Study IDs: Sentinel - 001
Record Dates: First submitted 2022-03-18; First posted 2022-03-31 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-03

CONDITIONS: Breathlessness; COPD; Asthma; Asthma Chronic; Wheezing; Dyspnea; Shortness of Breath
Keywords: Breathlessness; COPD; Asthma; Asthma Chronic; Wheezing; Dyspnea; Shortness of Breath
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe Breathlessness: Breathlessness requiring admission or supplementary oxygen
  Interventions: Other: Biomarker tests for participant profiling
- Moderate Breathlessness: Breathlessness requiring medical intervention < 24 hours without meeting the criteria for severe breathlessness
  Interventions: Other: Biomarker tests for participant profiling
- Mild Breathlessness: Breathlessness not requiring any medical intervention within 24 hours other than a dose change in the individuals pre-established pharmacological treatment plan
  Interventions: Other: Biomarker tests for participant profiling

INTERVENTIONS:
Other: Biomarker tests for participant profiling — Combination of digital and physical tests to objectify measures relevant for breathlessness

SUMMARY:
The Sentinel-001 study aims to identify a combination of biomarkers suitable for triage of breathlessness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90 years.
* Has experienced episode of breathlessness during the past 12 months triggering interaction with a health care professional. Self-reported breathlessness using any of the following words to describe symptoms will qualify as a presentation of breathlessness regardless of aetiology or severity of symptoms: shortness of breath, tight chest, trouble breathing, breathlessness, dyspnoeic, breathless, asthmatic, suffocating, wheezing, fighting for breath or any equivalent word. Breathlessness does not have to be the primary presenting symptom.
* Deemed clinically sufficiently stable to participate according to health care practitioner.

Exclusion Criteria:

* Inability to understand written local language at a year 5 level.
* Not being confident in use of digital technology (smartphone and/or tablet). This will become evident through an inability to use the system.
* Inability to enter required study sample data due to diminished consciousness and/or physical or mental capacity regardless of whether this is associated with the breathlessness event.
* Received an investigational medical product in the context of a Clinical Trial during the 28 days prior to first probe administration.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants having experienced episode of breathlessness during the past 12 months triggering interaction with a health care professional.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Physician assessed severity of breathlessness | 1 day (One-time assessment during a participant reported episode of breathlessness)
  Breathlessness requiring admission or supplementary oxygen, breathlessness requiring intervention < 24 hours, Breathlessness requiring medical intervention within 24 hours without meeting the criteria for severe breathlessness, Breathlessness not requiring any medical intervention within 24 hours other than a dose change in the individuals pre-established pharmacological treatment plan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith AK, Currow DC, Abernethy AP, Johnson MJ, Miao Y, Boscardin WJ, Ritchie CS. Prevalence and Outcomes of Breathlessness in Older Adults: A National Population Study. J Am Geriatr Soc. 2016 Oct;64(10):2035-2041. doi: 10.1111/jgs.14313. Epub 2016 Sep 7. PMID 27603500
- [Background] Tobin MJ, Laghi F, Jubran A. Why COVID-19 Silent Hypoxemia Is Baffling to Physicians. Am J Respir Crit Care Med. 2020 Aug 1;202(3):356-360. doi: 10.1164/rccm.202006-2157CP. PMID 32539537
- [Background] Barnes N, Calverley PM, Kaplan A, Rabe KF. Chronic obstructive pulmonary disease and exacerbations: patient insights from the global Hidden Depths of COPD survey. BMC Pulm Med. 2013 Aug 23;13:54. doi: 10.1186/1471-2466-13-54. PMID 23971625
- [Background] Coutinho AD, Lokhandwala T, Boggs RL, Dalal AA, Landsman-Blumberg PB, Priest J, Stempel DA. Prompt initiation of maintenance treatment following a COPD exacerbation: outcomes in a large insured population. Int J Chron Obstruct Pulmon Dis. 2016 Jun 8;11:1223-31. doi: 10.2147/COPD.S102570. eCollection 2016. PMID 27354781
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig LM, Moher D, Rennie D, de Vet HC, Lijmer JG; Standards for Reporting of Diagnostic Accuracy. The STARD statement for reporting studies of diagnostic accuracy: explanation and elaboration. Ann Intern Med. 2003 Jan 7;138(1):W1-12. doi: 10.7326/0003-4819-138-1-200301070-00012-w1. PMID 12513067
- See also: Health Research Authority. Is my study research? — http://www.hra-decisiontools.org.uk/research/
- See also: MHRA, Health and care research Wales, NHS Scotland, Health and Social Care & NHS Health Research Authority. Joint statement on seeking consent by electronic methods — https://s3.eu-west-2.amazonaws.com/www.hra.nhs.uk/media/documents/hra-mhra-econsent-statement-sept-18.pdf